CLINICAL TRIAL: NCT04264754
Title: Characterization of Methylation Patterns in Hepatocellular Carcinoma
Status: Terminated | Type: Observational
Why Stopped: Sponsor prioritize other clinical projects over this study
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Liver-RND-001
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Cirrhosis
Keywords: Cirrhosis; Hepatocellular Carcinoma; Methylation; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases Group: Subjects who have already been diagnosed with liver cancer, however did not yet undergo any surgery, ablation, embolization or any other treatment for this cancerous lesion (including, but not limited to systemic therapies)
  Interventions: Procedure: Blood collection
- Control Group: Cancer free subjects with high risk to development HCC. High risk subjects include the following:
  1. Subjects with HCV (hepatitis C virus) and cirrhosis
  2. Subjects with HBV (hepatitis B virus) and cirrhosis
  3. Non-cirrhotic chronic HBV subjects at intermediate or high risk of HCC, according to EASL (European Association for the Study of the Liver) Clinical Practice Guidelines for the management of hepatocellular carcinoma
  4. Subjects with NAFLD (Non-Alcoholic Fatty Liver Disease) with cirrhosis
  5. Cirrhotic patients due to any other reasons, including alcohol disease
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — Peripheral blood will be collected via routine venipuncture procedure

SUMMARY:
This study is being performed as part of the development process of the Liver EpiCheck test which includes the identification of different methylation profiles in HCC (hepatocellular carcinoma) patients compare to cancer free control in blood samples

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study aimed to collect blood samples and de-identified clinical data from subjects diagnosed with HCC (cases arm) and subjects with high risk for HCC which are undergoing routine surveillance for HCC.

ELIGIBILITY:
Inclusion Criteria - Case Group:

* Age ≥ 22 years
* Subjects who are willing and able to provide written informed consent
* Subjects with confirmed diagnosis of HCC, naïve to tumor directed therapy

Exclusion Criteria - Case Group:

* Subjects with current cancer of any kind, other than hepatocellular carcinoma
* Subjects with a history of cancer of any kind (including hepatocellular carcinoma), other than non-melanoma skin cancer completely resected
* Coinfection with HIV
* Prior solid organ transplant

Inclusion Criteria - Control Group:

* Age ≥ 22 years
* Subjects who are willing and able to provide written informed consent
* Subjects diagnosed with one of the following:

  i. Subjects with HCV and cirrhosis ii. Subjects with HBV and cirrhosis iii. Non-cirrhotic chronic HBV subjects at intermediate or high risk of HCC, according to EASL Clinical Practice Guidelines for the management of hepatocellular carcinoma iv. Subjects with Non-Alcoholic Fatty Liver Disease (NAFLD) with cirrhosis. v. Cirrhotic patients due to any other reasons, including alcohol disease
* Subjects currently undergoing surveillance for hepatocellular carcinoma
* HCC surveillance imaging (e.g., US, CT, MRI) performed within 3 months prior to baseline visit
* Subjects with compensated liver function as measured by Child-Pugh Score A or B7 without ascites (all measures should be from the last three months)

Exclusion Criteria - Control Group:

* Subjects with current cancer of any kind, other than hepatocellular carcinoma
* Subjects with a history of cancer of any kind (including hepatocellular carcinoma), other than non-melanoma skin cancer completely resected
* Coinfection with HIV
* Prior solid organ transplant
* Current substance abuse

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have already been diagnosed with liver cancer, however did not yet undergo any surgery, ablation, embolization or any other treatment for this cancerous lesion (including, but not limited to systemic therapies) will be enlisted into the study as the Case group.
  In addition, blood samples will be obtained from participants without cancer, who are considered in high risk for HCC; those subjects will be recruited from outpatient units or from Health Management Organization involved in routine surveillance for HCC in high risk subjects.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
To collect blood samples and clinical data in order to characterize methylation patterns that will discriminate between HCC and normal hepatic tissue | 60 months
  To collect blood samples and clinical data in order to characterize methylation patterns that will discriminate between HCC and normal hepatic tissue
To develop a molecular blood test that will be able to detect HCC based on change in methylation patterns between HCC and normal hepatic tissue | 60 months
  To develop a molecular blood test that will be able to detect HCC based on change in methylation patterns between HCC and normal hepatic tissue

SECONDARY OUTCOMES:
Liver EpiCheck Performance | 60 months
  To assess the performance of the Liver EpiCheck in terms of (1) Sensitivity (2) Specificity (3) NPV(negative predictive value) and (4) PPV (positive predictive value)

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - Ha'emek Medical Center, Afula
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
No IPD will be share with other researchers. The statistical analysis will be performed by the study sponsor